CLINICAL TRIAL: NCT05611905
Title: Phase 1 Biodistribution and Pathophysiology Study of 11C-para-aminobenzoic Acid (11C-PABA)
Brief Title: Biodistribution and Pathophysiology Study of 11C-para-aminobenzoic Acid
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00179210; R01HL131829 (NIH)
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Renal Excretion; Bacterial Infections; Inflammatory Disease; Oncologic Disease
Keywords: PET/CT; Probenecid; 11C-PABA
MeSH Terms: conditions — Bacterial Infections | interventions — Probenecid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 11C-para-aminobenzoic acid PET/CT
  Interventions: Combination Product: 11C-para-aminobenzoic acid PET/CT; Drug: Probenecid

INTERVENTIONS:
Combination Product: 11C-para-aminobenzoic acid PET/CT — A bolus of 20 mCi of 11C-PABA followed by PET/CT
Drug: Probenecid — Oral dose of 500 mg (tablet) 2 hours before IV dose of 11C-PABA will be administered.

SUMMARY:
The investigators will perform radionuclide PET scans in subjects with infectious diseases to assess whether radio-labeled PABA (11C-PABA) is effective for infection imaging.

Tomographic imaging can be used to evaluate disease processes deep within the body, noninvasively and relatively rapidly. The goal is to see if this imaging technique can help differentiate infections from non-infectious processes and also provide information on the causative bacterial class.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age at the time of consent and imaging.
2. Healthy subjects OR those with confirmed (microbiologically, molecular or serological testing) diagnosis of infection at any body site OR clinical and imaging evidence of suspected infection in any body site with confirmation (microbiologically, molecular or serological testing) anticipated within 72 hours of imaging.

   OR subjects with confirmed inflammatory (rheumatoid arthritis, idiopathic pulmonary fibrosis, etc) or oncologic (e.g. localized or metastatic tumors) disease and clinically determined not to have infection.
3. For subjects with infections:

   Non mycobacterium tuberculosis infections: received no more than 7 days of effective antibiotic treatment, as judged by the attending and/or principal investigator.

   OR Mycobacterium tuberculosis or mycobacteroides infections: received no more than 4 weeks of effective treatment. Infection confirmed by positive culture or molecular testing.
4. For inpatients, determined by the attending of record to be stable to participate in the study (will be documented in the research records).
5. Subject is judged by the investigator to have the initiative and means to be compliant with the protocol.
6. Subjects or their legal representatives must have the ability to read, understand and provide written informed consent for the initiation of any study related procedures. Adults lacking capacity will not be enrolled in this study.

Exclusion criteria:

Within 28 or fewer days prior to imaging, a complete blood count with differential, blood comprehensive metabolic panel will be performed. Subjects will be excluded from enrollment if any of the following apply:

1. Reported pregnancy or pregnancy as determined by positive or indeterminate serum human chorionic gonadotrophin (hCG) at screening and positive urine hCG prior to radiopharmaceutical dosing.
2. Lactating females.
3. Inadequate venous access.
4. Screening clinical laboratory values must be within normal limits or judged not clinically significant by the principal investigator.
5. Administered a radioisotope within 5 physical half-lives prior to study enrollment.
6. Subject has been treated with an investigational drug / biologic / therapeutic device within 30 days prior to study radiotracer administration.
7. Determined to have prior (external) radiation exposure which will exceed RDRC annual radiation exposure limit of 5 rems.
8. For patients undergoing renal imaging they will be excluded if any of the following conditions exist:

   * Hypertension
   * Diabetes mellitus type I or II
   * Body mass index less than 18.5 kg/m2 or higher than 30 kg/m2
   * Family history of renal disease
   * Urinary tract infection in the prior 6 months

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with bacterial infections or non-infectious processes such as inflammatory / oncologic diseases will be enrolled. Males and female members of all races and ethnic groups are eligible for this trial and encouraged to participate.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-12-22 (Actual); Primary Completion 2025-11-08 (Actual); Study Completion 2025-11-08 (Actual)

PRIMARY OUTCOMES:
Pathophysiology of 11C-PABA in diseased subjects | Up to 3 hours
  Reconstruction of the PET data will be performed by means of iterative reconstruction (IR) by the ordered subset-expectation-maximization (OSEM) method with CT attenuation correction.
Biodistribution of 11C-PABA in diseased subjects | Up to 3 hours
  Reconstruction of the PET data will be performed by means of iterative reconstruction (IR) by the ordered subset-expectation-maximization (OSEM) method with CT attenuation correction.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay K Jain, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States